CLINICAL TRIAL: NCT02094560
Title: Phase II Trial of CAP7.1 in Adult Patients With Refractory Malignancies: Small Cell Lung Carcinoma, Non-Small Cell Lung Carcinoma, Biliary Carcinoma (PIITCAP)
Brief Title: CAP7.1 for the Treatment of Advanced Stage, Therapy Refractory Lung and Biliary Tract Tumors
Acronym: CAP7-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated to be redesigned for a trial according to EMA proposal.
Sponsor: CellAct Pharma GmbH (Industry)
Collaborators: Mundipharma-EDO GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPN710102; 2012-002378-30 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Advanced Endstage Solid Carcinomas in Adults
Keywords: therapy refractory; endstage; solid tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Small cell lung cancer (Experimental): Histologically- or cytologically-confirmed, limited and extensive SCLC disease with progression after first or second line treatment
  Interventions: Drug: CAP7.1
- Non small cell lung cancer (Experimental): Histologically- or cytologically-confirmed diagnosis of NSCLC with Stage IIIB or IV after failure of at least two lines of therapy
  Interventions: Drug: CAP7.1
- biliary tract cancer (Experimental): Histologically or cytologically confirmed diagnosis of biliary tract cancer progress after first line therapy
  Interventions: Drug: CAP7.1

INTERVENTIONS:
Drug: CAP7.1 — CAP7.1 is a prodrug of Etoposide released after via specific carboxyesterase

SUMMARY:
To assess the anti-tumor activity of CAP7.1 based on the observed objective response rate and rate of disease stabilization, as defined by the below primary and secondary endpoints, in patients with Non-Small Cell Lung Carcinoma (NSCLC), SCLC or biliary cancer who have progressed despite one or more previous chemotherapy line.

DETAILED DESCRIPTION:
A phase II evaluation will be performed in adult patients in parallel studies in 3 tumor types: NSCLC, SCLC and Biliary Tract Cancer. All patients will have advanced or metastatic disease with primary or secondary resistance to standard therapy. In each tumor type the patients will be randomized to receive either therapy with CAP7.1 or best supportive care according to institution standards. Patient in the Control group who progress may cross over to CAP7.1, however these patients will be analyzed separately from the patients randomized to CAP7.1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed, advanced disease with documented progression (RECIST1.1.) after one or several chemotherapy line
* Patients may also have received molecular targeted therapy and progressed while on therapy or after completion
* Must have recovered from the acute reversible effects of previous anti-cancer chemotherapy, usually 3-4 weeks after myelosuppressive chemotherapy

Exclusion Criteria:

* Serious concurrent medical condition, which could affect compliance with the protocol or interpretation of results.
* Patients with uncontrolled infection and patients known to be infected with the human immunodeficiency virus (HIV) or hepatitis infection are not eligible for the study
* Pregnancy or breast-feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11-08 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | 18 month
  Assessment of antitumor activity based on RECIST 1.1 criteria (complete response; partial response; stable disease)

SECONDARY OUTCOMES:
1. Percentage of Subjects With Objective Response [i.e., complete response (CR) + partial response (PR)] According to RECIST1.1 | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Time to Treatment Failure | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Progression-Free Survival (PFS) | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Disease-free survival | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Overall Survival (OS) | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Number of Subjects With Treatment Emergent Adverse Events (TEAEs) | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Maximum Observed Drug Concentration (Cmax) of CAP7.1 in Plasma | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Time to Reach Maximum Drug Concentration (tmax) of CAP7.1 in Plasma | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Half-life Associated With the Terminal Slope (t1/2) of CAP7.1 in Plasma | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)
Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC) of CAP7.1 in Plasma | Start of study treatment until 26 days post-last study treatment (approximately 4 years and 2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite, University Hospital, Berlin, Germany

REFERENCES:
- [Derived] Keilholz U, Rohde L, Mehlitz P, Knoedler M, Schmittel A, Kummerlen V, Klinghammer K, Treasure P, Lassus M, Steventon G, Machacek M, Utku N. First-in-man dose escalation and pharmacokinetic study of CAP7.1, a novel prodrug of etoposide, in adults with refractory solid tumours. Eur J Cancer. 2017 Jul;80:14-25. doi: 10.1016/j.ejca.2017.03.032. Epub 2017 May 19. PMID 28531881